CLINICAL TRIAL: NCT02449837
Title: Investigation of Circulating Tumor Cells From Cancer Patients Undergoing Radiation Therapy
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1408
Record Dates: First submitted 2015-04-07; First posted 2015-05-20 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Circulating Tumor Cells
MeSH Terms: conditions — Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (10):
- Head and Neck Cancer: Patient with locally advanced head and neck cancer but no distant metastasis scheduled to receive radiotherapy to the head and neck region with or without chemotherapy/targeted therapy (palliative or curative intent).
  Interventions: Other: Blood draw
- Cervical Cancer: Patients with locally advanced cervical cancer without distant metastasis scheduled for radiotherapy to the pelvic region with or without chemotherapy/targeted therapy (palliative or curative intent).
  Interventions: Other: Blood draw
- Non-Small Cell Lung Cancer: Patients with stage I to III non-small cell lung cancer, without distant metastasis, scheduled to receive stereotactic body radiotherapy for early stage lung disease and/or external beam radiotherapy for locally advanced lung disease, with or without concurrent/sequential chemotherapy and/or targeted therapy (curative intent).
  Interventions: Other: Blood draw
- Rectal Cancer: Patients with locally advanced rectal cancer (no distant metastasis) scheduled to receive neoadjuvant chemoradiotherapy (curative intent).
  Interventions: Other: Blood draw
- Metastatic Prostate Cancer: Patients with metastatic prostate cancer scheduled for palliative radiotherapy, or biochemically recurrent prostate cancer following radical prostatectomy scheduled for salvage prostatic fossa radiotherapy, with or without androgen deprivation, or with high risk prostate cancer.
  Interventions: Other: Blood draw
- Oligometastatic Disease: Patients with oligometastatic cancer, defined as any solid malignancy with< 5 measurable sites of metastatic disease, limited to a maximum of 3 anatomic organ systems, excluding the primary tumor and regional lymph nodes. At least 1 site of metastatic disease, but as many as all 5 sites, in addition to the primary tumor and regional lymph nodes, is amenable to local ablative therapy with external beam radiation, stereotactic cranial radiosurgery or stereotactic body radiotherapy. Treatment will be guided by multi-disciplinary evaluation and may also include surgery, chemotherapy or target agents at the discretion of the primary oncologists. Patients may present with oligometastatic disease or have oligometastatic disease recurrence after definitive therapy for localized disease.
  Interventions: Other: Blood draw
- Immunotherapy: Melanoma or metastatic NSCLC scheduled to receive ipilimumab, nivolumab, and/or pembrolizumab.
  Interventions: Other: Blood draw
- Head and Neck Induction chemotherapy: Locally advanced head and neck cancer (HNSCC) scheduled to receive induction chemotherapy followed by radiotherapy.
  Interventions: Other: Blood draw
- Metastatic Breast Cancer: Patients scheduled to receive any treatment, including radiation therapy, and/or systemic/hormonal therapy
  Interventions: Other: Blood draw
- Endometrial Cancer: Patients with stage III endometrial cancer, being treated with adjuvant radiation
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Blood samples will be collected at up to 4 time points before and during radiation. Blood will be collected at least 4 to 12 weeks post-treatment. Additional post-treatment blood draws will be performed at each subsequent follow-up visit to UNC (roughly ~1 month interval), up until 24 months after completion of radiation.

SUMMARY:
The purpose of this study is to investigate the level of Circulating Tumor Cells (CTCs) in cancer patients before and after undergoing treatment regimens where the primary treatment modality is radiation therapy (XRT). Specifically, there is interest in the change in CTCs pre- and post- XRT, both in absolute and relative terms.

DETAILED DESCRIPTION:
CTCs measurements will be taken pre- and post-RT treatment. CTCs measurements will also be taken during treatment. The CTCs measurements from this study will provide essential information for the power and sample size considerations for future translational studies, particularly for those looking to identify biomarkers possibly associated with CTCs and tumor response activity after XRT, and to adequately power more formal statistical comparisons of important associations between CTCs and patient characteristics and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cancer, fitting one of the following cohorts: locally advanced head and neck cancer but no distant metastasis scheduled to receive radiotherapy to the head and neck region with or without chemotherapy/targeted therapy (palliative or curative intent); locally advanced cervical cancer without distant metastasis scheduled for radiotherapy to the pelvic region with or without chemotherapy/targeted therapy (palliative or curative intent); Stage I to III non-small cell lung cancer, without distant metastasis, scheduled to receive stereotactic body radiotherapy for early stage lung disease and/or external beam radiotherapy for locally advanced lung disease, with or without concurrent/sequential chemotherapy and/or targeted therapy (curative intent); metastatic prostate cancer scheduled for palliative radiotherapy, or biochemically recurrent prostate cancer following radical prostatectomy; scheduled for salvage prostatic fossa radiotherapy, with or without androgen deprivation or with high risk prostate cancer; locally advanced rectal cancer (no distant metastasis) scheduled to receive neoadjuvant chemoradiotherapy (curative intent); oligometastatic cancer, defined as any solid malignancy with< 5 measurable sites of metastatic disease, limited to a maximum of 3 anatomic organ systems, excluding the primary tumor and regional lymph nodes. At least 1 site of metastatic disease, but as many as all 5 sites, in addition to the primary tumor and regional lymph nodes, is amenable to local ablative therapy with external beam radiation, stereotactic cranial radiosurgery (SRS) or stereotactic body radiotherapy (SBRT). Treatment will be guided by multi-disciplinary evaluation and may also include surgery, chemotherapy or target agents at the discretion of the primary oncologists. Patients may present with oligometastatic disease or have oligometastatic disease recurrence after definitive therapy for localized disease; Melanoma or metastatic NSCLC scheduled to receive ipilimumab, nivolumab, and/or pembrolizumab.; Locally advanced head and neck cancer (HNSCC) scheduled to receive induction chemotherapy followed by radiotherapy; Metastatic breast cancer scheduled to receive any treatment, including radiation therapy and/or systemic/hormonal therapy; Stage III endometrial cancer scheduled to receive radiation therapy
* Scheduled to initiate radiation for management of their disease, and schedule accommodates blood sample collection prior to radiation
* Male and female of ≥18 years of age
* Male and female patients capable of reproduction must agree to use medically acceptable methods of contraception, such as an intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence during radiation therapy. Inclusion of females of childbearing potential requires a negative pregnancy test within 14 days prior to study initiation (part of standard of care in radiation oncology).
* Written informed consent obtained and signed
* Able to have blood collection without excessive difficulty

Exclusion Criteria:

* Patient unwilling or unable to complete informed consent
* Physical or psychological inability to complete sample collection for any reason including but not limited to: inability to tolerate any study procedures, any physical limitation that would undermine the safety of the subject in the study, or any psychiatric or neurological condition that inhibits full comprehension of study requirements and inability to complete informed consent, as determined by treating physician
* Currently pregnant or lactating women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing radiation treatments at Lineberger Comprehensive Cancer Center at UNC Hospitals for one of eight cancer types: head and neck, cervical, rectal, lung, prostate, endometrial, metastatic breast, and oligometastatic cancer with any solid tumor histology. Additionally, patients undergoing immunotherapy at Lineberger Comprehensive Cancer Center at UNC Hosptials, or undergoing induction chemotherapy for treatment of head and neck cancers.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
To measure CTCs levels to evaluate the change pre- and post-treatment separately in 10 cohorts of patients receiving radiation therapy. | 24 months post-radiation

SECONDARY OUTCOMES:
Change in CTC levels from Baseline to Post-RT treatment and the correlation with local tumor response or pathological evaluation, depending on cohort | 24 months post-radiation

CONTACTS AND LOCATIONS:
Overall Officials: Dana Casey, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina, United States